CLINICAL TRIAL: NCT01846351
Title: Visual and Anatomic Outcomes of Intravitreal Anti-VEGF Therapy for Exudative Age-related Macular Degeneration With Concurrent Significant Epiretinal Membrane.
Brief Title: Intravitreal Anti-VEGF in Exudative AMD With Epiretinal Membranes
Status: Completed | Type: Observational
Sponsor: New England Retina Associates (Other)
Responsible Party: Principal Investigator, Peter E. Liggett, Principal Investigator, New England Retina Associates
Other Study IDs: NAC270608
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Epiretinal Membrane; Age Related Macular Degeneration
Keywords: choroidal neovascularization; epiretinal membrane; anti-VEGF
MeSH Terms: conditions — Epiretinal Membrane; Macular Degeneration; Choroidal Neovascularization

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Study designed to evaluate the effect of significant ERM on the visual and anatomic outcomes of intravitreal anti-VEGF therapy for eAMD.

DETAILED DESCRIPTION:
Gass in 1987 described three cases of epiretinal membrane (ERM) associated with wet macular degeneration. Since then we have seen that is not rare to find the coexistence of these entities. An ERM may produce intrinsic disorganization of the outer retina leading to persistent increased macular thickness and/or edema. This persistent edema may affect the effectiveness in the treatment of exudative age-related macular degeneration (eAMD). Therefore, this study was designed to evaluate the effect of significant ERM on the visual and anatomic outcomes of intravitreal anti-VEGF therapy for eAMD.

ELIGIBILITY:
Inclusion Criteria:

* Significant epiretinal membrane
* Anti-VEGF treatment for age-related macular degeneration

Exclusion Criteria:

* Uveitis
* Macular disorders
* Diabetic retinopathy
* Vascular occlusions

Ages: 58 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: age-related macular degeneration
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2006-07; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity | 12 months
  Evaluate the best visual acuity during the follow up.
Central macular thickness | 12 months
  Evaluation of the retinal thickness changes with anti-VEGF treatment
Fluorescein angiogram | 12 months
  Evaluation of changes in lesion size during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Nauman A Chaudhry, MD, Principal Investigator — New England Retina Associates; Peter E Liggett, MD, Study Chair — New England Retina Associates